CLINICAL TRIAL: NCT02746731
Title: Randomized Controlled Trial Assessing the Value of Prehabilitation in Patients Undergoing Colorectal Surgery According to the ERAS Protocol for the Improvement of Postoperative Outcomes
Brief Title: Prehabilitation - Enhanced Recovery After Colorectal Surgery
Acronym: pERACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Winterthur KSW (Other)
Collaborators: University of Zurich (Other); Zurich University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: pERACS
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Surgical Operation With Reversal of External Stoma; Colorectal Surgery
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prehabilitation (Experimental): 'Cardiorespiratory and resistance training.
  Interventions: Other: Cardiorespiratory and resistance training.
- Reference (Active Comparator): Usual care.
  Interventions: Other: Reference

INTERVENTIONS:
Other: Cardiorespiratory and resistance training. — A cardiorespiratory and resistance training program for at least 2 to 3 weeks will be conducted 3-times per week, of which two sessions will be supervised by a qualified person of the institute of physiotherapy and one session will be unsupervised and home-based.
  Physiotherapy consists of one hour, moderate to intense interval training combined with muscle strength training.
  Arms: Prehabilitation
Other: Reference — No preoperative physical therapy training. Patients will be informed to remain physically active (as usual) until surgery.
  Other Names: Usual care.
  Arms: Reference

SUMMARY:
The purpose of this study is to determine whether a combined cardiorespiratory and strengthening training prior to colorectal surgery decreases the rate of surgery-related complications.

DETAILED DESCRIPTION:
This single site study investigates whether a preoperative training reduces the number and severity of perioperative complications in patients undergoing elective colorectal surgery according to the Enhanced Recovery After Surgery (ERAS) pathway.

The study will be approved by a local ethical committee and conducted in compliance with the protocol, the current version of the Declaration of Helsinki, the ICH-GCP as well as all national legal and regulatory requirements. Before inclusion informed written consent will be obtained from all patients.

Once the indication for the surgical intervention is given patients may be included into the study. Patients of the experimental group will be provided with a tailored training program aiming at maximally improving physical fitness in order to withstand the surgical stress. Depending on the urgency of the operation this training program will last between two and six weeks. Three weekly trainings are foreseen of which two will be performed in a setting supervised by a physiotherapist and one at the patient's home.

Patients assigned to the control group receive the usual care i.e. information about the upcoming procedure and the advice to remain physically active.

From the point of the operation both groups will be treated equally. Outcome measures will be obtained from the inclusion into the study up to one month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years) suffering from colorectal diseases needing an operative treatment and treated along our ERAS pathway
* Patients suffering from colorectal cancer, diverticulosis, benign tumors such as polyps or inflammatory bowel disease and surgically treated (i.e. rectosigmoid resection, anterior resection of rectum, ileocaecal/right hemicolectomy, left hemicolectomy, abdominoperineal resection or total/subtotal colectomy), and patients undergoing reversal of Stoma and Hartmann procedures will be included.
* Informed Consent as documented by signature

Exclusion Criteria:

* Patients suffering from severe dementia or other cognitive impairment, what hinders them to give informed consent
* Patients with a physical impairment, who can't perform the necessary physical Training
* Patients, who are not able or willing to attend the physical training at the institute of physiotherapy of the Kantonsspital Winterthur
* Inability of the participant to follow the procedures of the study, e.g. due to language problems, psychological disorders, etc.
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-06; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Comprehensive Complication Index (CCI) | 30 days
  ssessment of patients' overall morbidity. CCI is based on the complication grading by Clavien-Dindo Classification and implements every occurred complication after an intervention. The overall morbidity is reflected on a scale from 0 (no complication) to 100 (death).

SECONDARY OUTCOMES:
Clavien/Dindo | 30 days
  Assessment of post-surgical complications, ranging from Grade I (any deviation from normal postoperative Course) to Grade V (death of Patient).
Five Times Sit to Stand Test | 30 days
  Time needed to raise from and sit-down on a chair for five times.
2-Minute Walk Test | 30 days
  Distance covered within two minutes of brisk walking.
Perceived pain | 30 days
  Numeric rating scale ranging from Zero (no pain) to ten (worst pain).

OTHER OUTCOMES:
The self-reported International Physical Activity Questionnaire short-form (IPAQ-SF) | 30 days
  The IPAQ is used as a comparable and standardised self-report measure of habitual physical activity.
hand grip strength | 30 days
  Jamar handheld dynamometer.
Rating of Perceived Exertion | 30 days
  Borg scale.
Steep ramp test | 30 days
  Test to determine training intensity.
Modified Iowa Levels of Assistance Scale (Milas) | 30 days
  Measure to quantify the gait and mobility impairments

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Breitenstein, MD, PD, Study Chair — Kantonsspital Winterthur KSW
Locations (1):
- Kantonsspital Winterthur, Winterthur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bardram L, Funch-Jensen P, Jensen P, Crawford ME, Kehlet H. Recovery after laparoscopic colonic surgery with epidural analgesia, and early oral nutrition and mobilisation. Lancet. 1995 Mar 25;345(8952):763-4. doi: 10.1016/s0140-6736(95)90643-6. PMID 7891489
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Dronkers JJ, Chorus AM, van Meeteren NL, Hopman-Rock M. The association of pre-operative physical fitness and physical activity with outcome after scheduled major abdominal surgery. Anaesthesia. 2013 Jan;68(1):67-73. doi: 10.1111/anae.12066. Epub 2012 Nov 5. PMID 23121372
- [Background] Slankamenac K, Graf R, Barkun J, Puhan MA, Clavien PA. The comprehensive complication index: a novel continuous scale to measure surgical morbidity. Ann Surg. 2013 Jul;258(1):1-7. doi: 10.1097/SLA.0b013e318296c732. PMID 23728278
- [Background] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, Macfie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery (ERAS) Society, for Perioperative Care; European Society for Clinical Nutrition and Metabolism (ESPEN); International Association for Surgical Metabolism and Nutrition (IASMEN). Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS((R))) Society recommendations. World J Surg. 2013 Feb;37(2):259-84. doi: 10.1007/s00268-012-1772-0. No abstract available. PMID 23052794
- [Derived] Gloor S, Misirlic M, Frei-Lanter C, Herzog P, Muller P, Schafli-Thurnherr J, Lamdark T, Schregel D, Wyss R, Unger I, Gisi D, Greco N, Mungo G, Wirz M, Raptis DA, Tschuor C, Breitenstein S. Prehabilitation in patients undergoing colorectal surgery fails to confer reduction in overall morbidity: results of a single-center, blinded, randomized controlled trial. Langenbecks Arch Surg. 2022 May;407(3):897-907. doi: 10.1007/s00423-022-02449-0. Epub 2022 Jan 27. PMID 35084526
- [Derived] Taha A, Taha-Mehlitz S, Staartjes VE, Lunger F, Gloor S, Unger I, Mungo G, Tschuor C, Breitenstein S, Gingert C. Association of a prehabilitation program with anxiety and depression before colorectal surgery: a post hoc analysis of the pERACS randomized controlled trial. Langenbecks Arch Surg. 2021 Aug;406(5):1553-1561. doi: 10.1007/s00423-021-02158-0. Epub 2021 Mar 29. PMID 33782738
- [Derived] Merki-Kunzli C, Kerstan-Huber M, Switalla D, Gisi D, Raptis DA, Greco N, Mungo G, Wirz M, Gloor S, Misirlic M, Breitenstein S, Tschuor C. Assessing the Value of Prehabilitation in Patients Undergoing Colorectal Surgery According to the Enhanced Recovery After Surgery (ERAS) Pathway for the Improvement of Postoperative Outcomes: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2017 Oct 27;6(10):e199. doi: 10.2196/resprot.7972. PMID 29079551